CLINICAL TRIAL: NCT06095193
Title: The Effect of Education Applied to Women in Menopause on the Daily Effects of Vaginal Aging, Avoidance of Sexuality and Sexual Stress
Brief Title: The Effect of Education on Vaginal Effects of Menopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Ayşe Elkoca, Asist.Prof.Dr., Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GaziantepIslamSTU
Record Dates: First submitted 2023-10-05; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Menopause; Aging; Failure of Genital Response

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: menopause education (Experimental): Women will be taught the physiology of female reproductive organs, physiology of menopause, vaginal symptoms in menopause, sexual myths in menopause and practices that will support sexuality in menopause, in 50 minutes for 4 weeks.
  Interventions: Behavioral: menopause education
- control group (No Intervention): No intervention will be made

INTERVENTIONS:
Behavioral: menopause education — Women will be taught the physiology of female reproductive organs, physiology of menopause, vaginal symptoms in menopause, sexual myths in menopause and practices that will support sexuality in menopause, in 50 minutes for 4 weeks.
  Arms: Experimental: menopause education

SUMMARY:
The aim of our study is to examine the effect of education applied to women in menopause on the daily effects of vaginal aging, avoidance of sexuality and sexual stress. It is a pretest-posttest randomized controlled experimental study. The universe of the research; It consisted of menopausal women over the age of 45 who attended courses at Özgecan Cultural Center and Binevler Social Facility in Gaziantep. The sample of the research consisted of 102 people determined by the GPower method and determined by simple random method among all women who volunteered to participate in the study. Introductory Information Form, Daily Effect of Vaginal Aging Scale, Sexuality Avoidance Decision Balance Scale and Sexuality Avoidance Self-Efficacy Scale, Female Sexual Distress Scale were used to collect the research data. . The data will be collected face to face with the form prepared by the researchers after mass announcements and explanations are made to the women.

DETAILED DESCRIPTION:
Menopause is an inevitable event in every woman's life. This is a period in which women adapt to physical, emotional, mental and hormonal changes in their lives. During this process, the woman's menstrual cycle is permanently interrupted. The aim of our study is to examine the effect of education applied to women in menopause on the daily effects of vaginal aging, avoidance of sexuality and sexual stress. It is a pretest-posttest randomized controlled experimental study. This research was conducted between October 2023 and December 2023 with menopausal women over the age of 45 who attended courses at Özgecan Cultural Center and Binevler Social Facility in Gaziantep. The universe of the research; It consisted of menopausal women over the age of 45 who attended courses at Özgecan Cultural Center and Binevler Social Facility in Gaziantep. The sample of the research consisted of 102 people determined by the GPower method and determined by simple random method among all women who volunteered to participate in the study. Introductory Information Form, Daily Effect of Vaginal Aging Scale, Sexuality Avoidance Decision Balance Scale and Sexual Avoidance Self-Efficacy Scale, Female Sexual Distress Scale were used to collect the research data. . The data will be collected face to face with the form prepared by the researchers after mass announcements and explanations are made to the women.

ELIGIBILITY:
Inclusion Criteria:

* Being able to understand what you read
* being in menopause
* continue throughout education
* Being 45 years or older

Exclusion Criteria:

* being under 45
* having a mental problem
* not being in menopause
* not attending one of the training sessions

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-10-25 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of menopause education | 6 week
  Improvement in women's symptoms as a result of training

SECONDARY OUTCOMES:
Scale-1 | one week and last week
  DAILY IMPACT OF VAGINAL AGING SCALE
Scale-2 | one week and last week
  Female Sexual Distress Scale

IPD SHARING:
Plan to Share IPD: No
Indicate if there is a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Elkoca A, Ayar D. Effects of education given in the menopausal period on the day-to-day impact of vaginal aging, self-efficacy in sexual abstinence and sexual distress: A randomized clinical trial. Women Health. 2025 Jan;65(1):4-18. doi: 10.1080/03630242.2024.2432934. Epub 2024 Dec 1. PMID 39617952